CLINICAL TRIAL: NCT04440059
Title: A Multicenter, Open Clinical Trial to Evaluate the Safety and Efficacy of ICP-022 in the Treatment of Recurrent or Refractory Waldenstrom Macroglobulinemia (WM)
Brief Title: A Study of ICP-022 in the Treatment of Recurrent or Refractory Waldenstrom Macroglobulinemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-00105
Record Dates: First submitted 2020-06-16; First posted 2020-06-19 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Waldenstrom's Macroglobulinemia Recurrent; Waldenstrom's Macroglobulinemia Refractory

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICP-022 (Experimental): Subjects will take ICP-022 150mg once daily (QD).
  Interventions: Drug: ICP-022

INTERVENTIONS:
Drug: ICP-022 — ICP-022 at a dose of 150mg PO QD

SUMMARY:
The phase II clinical study is to investigate the safety, tolerability, efficacy and pharmacokinetics of ICP-022.

Safety, tolerability evaluation, and anti-tumor effects of ICP-022 in Chinese patients with R/R WM will be evaluated in approximately 44 subjects. Pharmacokinetics of ICP-022 will be evaluated in approximately 20 subjects.

ELIGIBILITY:
Key Inclusion criteria:

1. Clinical and histologically confirmed giant globulinemia Fahrenheit (WM Ii International Working Group Standards, IWWM-2, 2003) (Owen et al., 2003)
2. At least one treatment indication is met (7th WM International Working Group standards, IWWM-7) (Dimopoulos et al., 2014)
3. With the lowest serum IgM value >2 times ULN as the efficacy evaluation index
4. ECOG physical strength score 0-2
5. Voluntary written informed consent prior to trial screening.

Key Exclusion Criteria:

1. Present or prior history of other malignant neoplasms, unless radical treatment has been performed and there is no evidence of recurrence or metastasis in the last 5 years
2. Amyloidosis and central nervous system (CNS) involvement caused by WM
3. Demonstrate disease transformation
4. Patients who had received autologous stem cell transplantation within the previous 6 months
5. A history of organ transplantation or allogeneic bone marrow transplantation

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-08-10 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Major response rate（MRR） | Up to 3 years

SECONDARY OUTCOMES:
The occurrence of adverse events and serious adverse events | Cycle 1 (every 2 weeks), cycle 2-12 (every 4 weeks); After cycle 12 (every 12 weeks). Each cycle is 28 days.
  The safety of ICP-022 measured by the occurrence of adverse events and serious adverse events according to NCI-CTCAE 4.03 grading criteria
Duration of Major Mitigation (DOMR) | Evaluate during the screening period, 1-6 treatment cycle every 2 cycles (8 weeks), 6th-27th cycles every 3 cycles, evaluating every 6 cycles after the 27th cycle. Each cycle is 28 days.
Progression Free Survival (PFS) | Evaluate during the screening period, 1-6 treatment cycle every 2 cycles (8 weeks), 6th-27th cycles every 3 cycles, evaluating every 6 cycles after the 27th cycle. Each cycle is 28 days.

CONTACTS AND LOCATIONS:
Locations (16):
- China (16):
  - The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital), Hefei, Anhui
  - Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - West China hospital of sichuan university, Sichuan, Chengdu
  - Union Hospital affiliated to Fujian Medical University, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan Provincial Peoples's Hospital, Zhengzhou, Henan
  - Tongji Hospital affiliated to Huazhong University of Science and Technology, Wuhan, Hubei
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Ruijin Hospital affiliated to Shanghai Jiao Tong University, Shanghai, Shanghai Municipality
  - Hospital of Hematology, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - Union Hospital affiliated to Huazhong University of Science and Technology, Hubei, Wuhan
  - The First Affiliated Hospital of Zhejiang University Medical College, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Alfaifi A, Bahashwan S, Alsaadi M, Ageel AH, Ahmed HH, Fatima K, Malhan H, Qadri I, Almehdar H. Advancements in B-Cell Non-Hodgkin's Lymphoma: From Signaling Pathways to Targeted Therapies. Adv Hematol. 2024 Nov 12;2024:5948170. doi: 10.1155/2024/5948170. eCollection 2024. PMID 39563886
- [Derived] Cao XX, Jin J, Fu CC, Yi SH, Zhao WL, Sun ZM, Yang W, Li DJ, Cui GH, Hu JD, Liu T, Song YP, Xu B, Zhu ZM, Xu W, Zhang MZ, Tian YM, Zhang B, Zhao RB, Zhou DB. Evaluation of orelabrutinib monotherapy in patients with relapsed or refractory Waldenstrom's macroglobulinemia in a single-arm, multicenter, open-label, phase 2 study. EClinicalMedicine. 2022 Oct 4;52:101682. doi: 10.1016/j.eclinm.2022.101682. eCollection 2022 Oct. PMID 36313145